CLINICAL TRIAL: NCT03332875
Title: OurRelationship.Com Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Brian Doss, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140405
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Marital Conflict; Relationship, Marital
Keywords: OurRelationship; Couple therapy; Internet; Marriage Counseling

STUDY DESIGN:
Intervention Model Description: Couples are randomized to receive either one call with a coach or four calls with a coach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OurRelationship - 1 Coach Call (Experimental): OurRelationship online program plus a single call with a coach.
  Interventions: Behavioral: OurRelationship Online Program
- OurRelationship - 4 Coach Calls (Experimental): OurRelationship online program plus four calls with a coach.
  Interventions: Behavioral: OurRelationship Online Program

INTERVENTIONS:
Behavioral: OurRelationship Online Program — OurRelationship.com is an online program designed to improve distressed romantic relationships.

SUMMARY:
The purpose this study is to determine the continued reach and effectiveness of the OurRelationship.com program once paid advertising and payment for participation ceases. The answer to this question is essential to determining the sustainability of web-based interventions for couples. Specifically, this study has four aims:

1. Examine continued level of initial interest in the study, as measured by number of initial visits to the website, time spent on the page, and number of couples signing up for the study.
2. Measure any changes in the characteristics of the individuals expressing interest in the study, including demographics (e.g., race, ethnicity, education), relationship functioning (e.g., relationship satisfaction, previous help-seeking), and individual functioning (e.g., depression, anxiety)
3. Determine completion rates and effectiveness of the program once payments for participation have been removed.
4. Determine whether having a single Skype/phone call with a coach (rather than the four calls that were used in the NIH trial) significantly degrades completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a heterosexual relationship
* Married, Engaged, or living with partner for 6 months or more
* Living in the United States
* Both partners score at least 0.5 standards below the community mean on relationship satisfaction

Exclusion Criteria:

* Clinically significant intimate partner violence
* Younger than 18 or older than 64 years of age
* Reporting infidelity in last three months
* Reporting severe suicidal ideation in last three months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 712 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Relationship satisfaction | Change between baseline and the end of the intervention (approx. 2 months later)
  Relationship satisfaction as measured by the Couple Satisfaction Inventory, 16-item (Funk & Rogge, 2007; http://dx.doi.org/10.1037/0893-3200.21.4.572). Higher scores on this scale indicate greater satisfaction. Total scores range from 0 to 81, with a score below 51.5 indicating clinical distress. Internal consistency (alpha = 0.98) and convergent validity are strong.

SECONDARY OUTCOMES:
Depressive symptoms | Change between baseline and the end of the intervention (approx. 2 months later)
  Depressive symptoms as measured by the 10-item Center for Epidemiologic Studies Depression Scale (CES-D-10). Higher scores on this scale indicate greater depressive symptoms. The scale has been shown to have excellent sensitivity, specificity, and internal consistency (e.g., Irwin, Artin, & Oxman, 1999; doi:10.1001/archinte.159.15.1701).
Anxiety symptoms | Change between baseline and the end of the intervention (approx. 2 months later)
  Anxiety symptoms, as measured by the Generalized Anxiety Disorder Scale-7 (GAD-7; Spitzer, Kroenke, Williams, & Lowe; DOI: 10.1001/archinte.166.10.1092). Scores on this measure range from 0 to 21, with higher scores indicating greater anxiety symptoms. Sensitivity (89%), specificity (82%), and criterion validity are excellent for this measure.

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data available to qualified professionals.

REFERENCES:
- [Derived] Roddy MK, Rothman K, Doss BD. A randomized controlled trial of different levels of coach support in an online intervention for relationship distress. Behav Res Ther. 2018 Nov;110:47-54. doi: 10.1016/j.brat.2018.09.002. Epub 2018 Sep 13. PMID 30240874